CLINICAL TRIAL: NCT01305057
Title: Human Use Test on Skin Hydration and Skin Barrier Function
Brief Title: Efficacy Test on Skin Hydration and Skin Barrier Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmos Technical Center (Industry)
Collaborators: University of Dundee (Other)
Responsible Party: Hitoshi Masaki, Cosmos Technical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Cosmos1; hydration-1 (Other: Cosmos Technical Center)
Record Dates: First submitted 2011-01-13; First posted 2011-02-28 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: Dry Skin
Keywords: dry skin condition

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Evaluation of P-IP on hydration and barrier function (Experimental): Effects of P-IP on improvement of skin hydration and TEWL were examined.
  Interventions: Other: Pyridoxine tri-isopalmitate

INTERVENTIONS:
Other: Pyridoxine tri-isopalmitate — 2% dosage, oil-in-water emulsion, twice a day, 28 days

SUMMARY:
The effects of topically applied pyridoxine tri-isopalmitate (P-IP) which stimulates filaggrin synthesis in keratinocytes, on skin hydration and barrier function were examined. Subjects were separated into two groups to examine the effect of P-IP. Subjects were treated with P-IP formulation on one side of the face and with a placebo formulation on the other side twice daily (morning and evening) for 28 days. All subjects gave written informed consent prior to the study. The skin hydration and TEWL (transepidermal water loss) were evaluated by measuring skin surface conductance with a skin hygrometer SKICON 200EX (I.B.S. ltd., Japan) and TEWL meter AS-CT1 (ASAHI BIOMED, Tokyo, Japan), respectively.

DETAILED DESCRIPTION:
It is expected that the long-term application of P-IP increase skin surface water contents and suppress TEWL.

ELIGIBILITY:
Inclusion Criteria:

* healthy skin

Exclusion Criteria:

* don't use any moisturizer

Ages: 33 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Measurement of skin surface water content and Trans-Epidermal Water Loss (TEWL) | Before application, 1 week, 2 week and 4 weeks after application
  Subjects were treated with P-IP formulation on one side of the face and with a placebo formulation (without P-IP, oil-in-water emulsion type) on the other side twice daily (morning and evening) for 28 days. Skin surface water contents and TEWLs were measured at the time frame described above and the results were analyzed as a change from a value of before-application at each measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Cosmos Technical Center, Itabashi-ku, Tokyo, Japan